CLINICAL TRIAL: NCT02169804
Title: An Open-Label Study to Evaluate the Effect of Age Upon the Pharmacokinetics of Androxal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZA-111
Record Dates: First submitted 2014-06-16; First posted 2014-06-23 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Enclomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 70 years or older (Experimental): Non-smoking healthy adult males >or equal to 70 years of age.
  Interventions: Drug: Androxal 25 mg
- Under 60 years of age (Experimental): Non-smoking healthy adult males<60 years of age.
  Interventions: Drug: Androxal 25 mg

INTERVENTIONS:
Drug: Androxal 25 mg

SUMMARY:
• To determine and compare the pharmacokinetics (PK) of 3 doses of 25 mg Androxal in elderly healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Speak, read, and understand English or Spanish and is willing and able to provide written informed consent on an IRB-approved form prior to the initiation of any study procedures;
2. Male; age <60 or ≥70 years of age
3. No significant abnormal findings at the screening physical examination as evaluated by the Investigator;
4. Normal laboratory values (or abnormal but not clinically significant) at screening as determined by the Investigator;
5. Subject is willing to remain in the clinic for the screening visit and one overnight treatment visit after the 3rd dose of Androxal (approximately 36 hours for the treatment visit)
6. Must be able to swallow gelatin capsules

Exclusion Criteria:

1. Known hypersensitivity to Clomid;
2. Abnormal screening visit vital signs or clinical laboratory evaluation considered clinically significant by the Investigator;
3. A hematocrit >54% or a hemoglobin >17 g/dL.
4. Subject with a significant organ abnormality or disease as determined by the Investigator;
5. Any medical condition that would interfere with the study as determined by the Investigator;
6. Participation in a clinical trial with investigational medication within 30 days prior to study medication administration;
7. An acute illness within 5 days of study medication administration;
8. Positive urine drug screen at the screening visit;
9. Known history of HIV and/or Hepatitis B or C
10. Tobacco (nicotine products) use in the 3 months prior to the study;
11. A mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study and/or evidence of an uncooperative attitude, as determined by the Investigator;
12. History of venous thromboembolic disease (e.g. deep vein thrombosis or pulmonary embolism);
13. History of myocardial infarction, unstable angina, symptomatic heart failure, ventricular dysrhythmia, or known history of QTc interval prolongation;
14. An employee or family member of an employee of the study site or the Sponsor;
15. Previous participation in a clinical study of Androxal.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - The Cmax will be calculated. | 4 days
Pharmacokinetics - The Tmax will be calculated. | 4 days
Pharmacokinetics - The AUC0-24 will be calculated. | 4 days
Pharmacokinetics - the AUC0-∞ will be calculated. | 4 days
Pharmacokinetics - The t½ will be calculated. | 4 days

SECONDARY OUTCOMES:
Safety - Incidence of adverse events | 4 days
Safety -Mean change from baseline in laboratory values | 4 days
Safety - Mean change from baseline in vital signs | 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Miami, Florida, United States